CLINICAL TRIAL: NCT01834248
Title: A Phase I Study of DEC205mAb-NY-ESO-1 Fusion Protein (CDX-1401) Given With Adjuvant PoIylCLC in Conjunction With 5-Aza-2'Deoxycytidine (Decitabine) in Patients With MDS or Low Blast Count AML
Brief Title: DEC-205/NY-ESO-1 Fusion Protein CDX-1401and Decitabine in Treating Patients With Myelodysplastic Syndrome or Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 227712; NCI-2013-00565 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 227712 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2013-04-12; First posted 2013-04-17 (Estimated); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Acute Myeloid Leukemia; Alkylating Agent-Related Acute Myeloid Leukemia; Chronic Myelomonocytic Leukemia; Myelodysplastic Syndrome; Refractory Anemia With Excess Blasts in Transformation
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes | interventions — Decitabine; Injections; poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (CDX-1401, Poly ICLC, decitabine) (Experimental): Patients receive DEC-205/NY-ESO-1 fusion protein CDX-1401 SC and ID and poly-ICLC SC on days -14 and 15 of course 1 and on day 15 for courses 2-4. Patients also receive decitabine IV over 1 hour on days 1-5. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: DEC-205/NY-ESO-1 Fusion Protein CDX-1401; Drug: Decitabine; Other: Laboratory Biomarker Analysis; Drug: Poly ICLC

INTERVENTIONS:
Biological: DEC-205/NY-ESO-1 Fusion Protein CDX-1401 — Given SC and ID
  Other Names: CDX-1401
Drug: Decitabine — Given IV
  Other Names: 5-Aza-2'-deoxycytidine; Dacogen; Decitabine for Injection; Deoxyazacytidine; Dezocitidine
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Poly ICLC — Given SC
  Other Names: Hiltonol; Poly I:Poly C with Poly-L-Lysine Stabilizer; poly-ICLC; PolyI:PolyC with Poly-L-Lysine Stabilizer; Polyinosinic-Polycytidylic Acid Stabilized with Polylysine and Carboxymethylcellulose; Polyriboinosinic-Polyribocytidylic Acid-Polylysine Carboxymethylcellulose; Stabilized Polyriboinosinic/Polyribocytidylic Acid

SUMMARY:
This phase I trial studies the side effects and immune response to DEC-205/NY-ESO-1 fusion protein CDX-1401 and decitabine in patients with myelodysplastic syndrome or acute myeloid leukemia. DEC-205-NY-ESO-1 fusion protein, called CDX-1401, is a full length NY-ESO-1 protein sequence fused to a monoclonal antibody against DEC-205, a surface marker present on many immune stimulatory cells. This drug is given with another substance called PolyICLC, which acts to provoke any immune stimulatory cells which encounter the NY-ESO-1-DEC-205 fusion protein to produce an immune response signal against NY-ESO-1. Immune cells which have thus been primed to react against NY-ESO-1 may then attack myelodysplastic or leukemic cells which express NY-ESO-1 after exposure to the drug decitabine. The chemotherapy drug decitabine is thought to act in several different ways, first, it may directly kill cancer cells, and secondly, the drug can cause cancer cells to re-express genes that are turned off by the cancer, including the gene for NY-ESO-1. Giving DEC-205/NY-ESO-1 fusion protein (CDX-1401) and polyICLC together with decitabine may allow the immune system to more effectively recognize cancer cells and kill them.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the safety of Anti-DEC-205-NY-ESOI (CDX-1401) fusion protein (DEC-205/NY-ESO-1 fusion protein CDX-1401) given in combination with decitabine 20 mg/m^2 intravenously.

SECONDARY OBJECTIVES:

I. To evaluate NY-ESO-1 specific cellular and humoral immunity by determination of NY-ESO-1 specific antibody, and T-cell clones following standard treatment with 5-aza-2'-deoxycytidine (decitabine) in conjunction with immune sensitization with Anti-DEC 205-NY-ESO-I fusion protein (CDX-1401).

II. To determine the impact of decitabine treatment on peripheral blood cells from patients treated in this manner on NY-ESO-1 target gene expression, NY-ESO protein expression, NY-ESO-1 promoter methylation, and global deoxyribonucleic acid (DNA) methylation.

TERTIARY OBJECTIVES:

I. To record the response rate (complete response, partial response and hematological improvement) in myelodysplastic syndrome (MDS) or low blast count acute myeloid leukemia (AML) patients treated with the combination in order to provide descriptive characteristics.

OUTLINE:

Patients receive DEC-205/NY-ESO-1 fusion protein CDX-1401 subcutaneously (SC) and intradermally (ID) and poly-ICLC subcutaneously (SC) on days -14 and 15 of course 1 and on day 15 for courses 2-4. Patients also receive decitabine intravenously (IV) over 1 hour on days 1-5. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30, 60, 90, and 180 days.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a confirmed diagnosis of:

  * International Prognostic Scoring System (IPSS) intermediate-I, interrnediate-2 or high-risk MDS including chronic myelomonocytic leukemia (CMML) or
  * Low blast count AML with =< 30% blasts previously classified as refractory anemia with excess blasts in transformation who have not been previously treated with a hypomethylating agent
  * Patients with IPSS intermediate-1 disease with an isolated deletion of chromosome 5q must have previously failed treatment with lenalidomide
* Subjects with Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Total bilirubin =< 2 x upper limit of normal (ULN)
* Aspartate transaminase (AST/serum glutamic oxaloacetic transaminase [SGOT]) and alanine transaminase (ALT/serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN
* Serum creatinine =< 1.5 x ULN
* Any human leukocyte antigen (HLA) type
* Subjects of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 6 months after the last treatment; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Subject or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Subjects with life-threatening illnesses other than MDS, uncontrolled medical conditions or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, or put the study outcomes at risk
* AML associated with inv(16); t(16;16); t(8;21) or t(15;17)
* Subjects with uncontrolled or symptomatic arrhythmias, or any class 3 or 4 cardiac disease as defined by the New York Heart Association functional classification
* Subjects with symptomatic central nervous system (CNS) disease which is not adequately controlled
* Subjects who have received prior radiation therapy for extramedullary disease within 2 weeks of first dose
* Subjects with human immunodeficiency virus (HIV) or active infection with hepatitis C virus (HCV) or hepatitis B virus (HBV)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Subjects who are being treated with systemic corticosteroids
* Subjects who have hypersensitivity to decitabine
* History of auto-immune disease (e.g. thyroiditis, lupus) except vitiligo
* Pregnant or nursing female subjects
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the subject an unsuitable candidate to receive study drug
* Received an investigational agent within 30 days prior to enrollment
* Active malignancy with the exception of basal cell carcinoma, non-melanoma skin cancer, cervical carcinoma-in-situ; other prior malignancies in remission for less than 1 year
* Subjects previously treated with an allogeneic stem cell transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-07-30 (Actual); Primary Completion 2015-06-09 (Actual); Study Completion 2016-03-21 (Actual)

PRIMARY OUTCOMES:
Incidence of toxicity graded according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 30 days after last dose of study treatment
  Toxicity rates will be described using upper one-sided 95% Clopper Pearson binomial confidence intervals.

SECONDARY OUTCOMES:
Change in immune and molecular epigenetic response | Baseline to up to 16 weeks
  Summarized by descriptive statistics (means, medians, quartiles, etc.) Confidence intervals will be constructed for the median and the mean. Exploratory graphical analysis will be used to discover associations among variables. The statistical significance of the change in marker values resulting from treatment will be assessed using the (paired sample) Wilcoxon Signed Rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Griffiths, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States